CLINICAL TRIAL: NCT01985386
Title: Iron Absorption Mechanism From a Slow Release Iron Capsule Using the Gastric Delivery System (Ferrous Sulfate)
Brief Title: Iron Absorption From GDS Capsules II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof., Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: EK 2013-N-05-2
Record Dates: First submitted 2013-10-31; First posted 2013-11-15 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Iron Deficiency
Keywords: Iron absorption; Slow release iron; Gastric delivery system; Iron deficiency
MeSH Terms: conditions — Iron Deficiencies | interventions — ferrous sulfate; Meals

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GDS (gastric delivery system), meal (Experimental): GDS capsule with meal
  Interventions: Dietary Supplement: GDS capsule with meal
- Ferrous sulfate, meal (Active Comparator): Ferrous sulfate with meal
  Interventions: Dietary Supplement: Ferrous sulfate with meal

INTERVENTIONS:
Dietary Supplement: GDS capsule with meal — GDS capsule with meal
  Arms: GDS (gastric delivery system), meal
Dietary Supplement: Ferrous sulfate with meal — Ferrous sulfate with meal
  Arms: Ferrous sulfate, meal

SUMMARY:
Slow release iron capsules containing ferrous sulfate have been designed based on the gastric delivery system. Iron absorption from those capsules administered with and without meals will be measured using stable iron isotopes.

ELIGIBILITY:
Inclusion Criteria:

* female,
* age 18-50 years,
* max. body weight 65 kg,
* serum ferritin < 30 µg/l

Exclusion Criteria:

* pregnancy,
* lactation,
* regular intake of medication,
* blood donation or significant blood losses over the past 4 months

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption | 2 weeks after test meal consumption

SECONDARY OUTCOMES:
Serum isotope appearance | 1, 2, 4 and 8 hours on days 1 and 8

OTHER OUTCOMES:
Serum non transferrin bound iron | 1, 2, 4 and 8 hours on days 1 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Aeberli, PhD, Principal Investigator — ETH Zurich (Switzerland)
Locations (1):
- Human Nutrition Laboratory, ETH Zurich, Zurich, Switzerland